CLINICAL TRIAL: NCT01415167
Title: Proleukin Observational Registry to Evaluate the Treatment Patterns and Clinical Response in Malignancy
Brief Title: PROCLAIM Registry to Evaluate the Treatment Patterns and Clinical Response in Malignancy
Status: Completed | Type: Observational
Sponsor: Prometheus Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: 10PLK13
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Metastatic Renal Cell Carcinoma; Metastatic Melanoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this registry is to collect information on patients who are receiving treatment with Proleukin in an organized way, and to learn more about patient care during and after treatment.

DETAILED DESCRIPTION:
The PROCLAIM Registry is a US-based, multicenter Registry designed to establish a high quality observational database of real-world clinical data on HD IL-2 when used to treat patients with mRCC, mM or other malignancies. The Registry will not, in any way, suggest changes in the treatment or management of the patients enrolled in the Registry. Therefore, physicians will continue to manage and treat patients according to standard of care and their own judgment.

The PROCLAIM Registry will start with a retrospective pilot data collection from a de-identified finite number of patient cases abstracted from their existing medical charts. The features collected will be identical to those planned for the prospective registry. The resulting database will be used to formulate hypotheses to be tested using the prospective registry database. Patients utilized in the retrospective analysis will be excluded from the prospective portion of the Registry.

In the prospective portion of the Registry, sites will enroll patients who are expected to start a course of HD IL-2 therapy. Once enrolled, the patient must receive at least one dose of HD IL-2 to remain in the Registry. Patients will be treated and followed according to the site's standard of care. This Registry will in no way induce changes in the management of individual patients. Clinical data features will be entered into an Electronic Data Capture (EDC) system, and organized into a registry database.

The data contained in the registry database will be observational data. The PROCLAIM Registry does not stipulate patient care, specific visits or interventions but merely surveys standardized parameters regarding HD IL-2 and associated therapies as they are applied by treatment centers. The collection of standard data over time permits the evaluation of trends in patient survival and subsequent therapy exposure. The database will be used to answer future queries formulated by researchers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Must have received at least one course of high dose IL-2 or Proleukin
* Signed informed consent form

Exclusion Criteria:

* Prior high dose IL-2 or Proleukin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients starting high dose IL-2 or Proleukin therapy are eligible to participate
Sampling Method: Non-Probability Sample
Enrollment: 1690 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
A source of observational data that can be used to report and query patient care patterns, clinical outcomes and trends from high dose IL-2 or Proleukin therapy in treating malignant melanoma, or renal cell carcinoma or other malignancies. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wong, MD, Study Chair — MD Anderson
Locations (45):
- United States (45):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Moores UCSD Cancer Center, La Jolla, California
  - USC Norris Cancer Center, Los Angeles, California
  - Southern California Permanente Medical Group, Riverside, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Mount Sinai Medical Center Comprehensive Cancer Center, Miami Beach, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Rush Pres St Lukes Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Oncology Specialists, SC, Park Ridge, Illinois
  - Indiana University Melvin and Bren Simon Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - The Baton Rouge Clinic, AMC, Baton Rouge, Louisiana
  - Johns Hopkins, Lutherville, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Midwest Cancer Center - Legacy, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Saint Luke's-Roosevelt Hospital Center, New York, New York
  - Columbia University/Herbert Irving Comprehensive Cancer Center, New York, New York
  - The Research Foundation for The State University of New York, Syracuse, New York
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - University Hospitals Siedman Cancer Center, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Saint Luke's Hospital and Health Network, Bethlehem, Pennsylvania
  - The Pennsylvania State University and The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hillman Cancer Research Pavilion, Div. of Medical Oncology, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
  - Wheaton Franciscan Cancer Care, Franklin, Wisconsin

REFERENCES:
- [Derived] Fishman M, Dutcher JP, Clark JI, Alva A, Miletello GP, Curti B, Agarwal N, Hauke R, Mahoney KM, Moon H, Treisman J, Tykodi SS, Daniels G, Morse MA, Wong MKK, Kaufman H, Gregory N, McDermott DF. Overall survival by clinical risk category for high dose interleukin-2 (HD IL-2) treated patients with metastatic renal cell cancer (mRCC): data from the PROCLAIMSM registry. J Immunother Cancer. 2019 Mar 27;7(1):84. doi: 10.1186/s40425-019-0567-3. PMID 30917871
- [Derived] Curti B, Daniels GA, McDermott DF, Clark JI, Kaufman HL, Logan TF, Singh J, Kaur M, Luna TL, Gregory N, Morse MA, Wong MKK, Dutcher JP. Improved survival and tumor control with Interleukin-2 is associated with the development of immune-related adverse events: data from the PROCLAIMSM registry. J Immunother Cancer. 2017 Dec 19;5(1):102. doi: 10.1186/s40425-017-0307-5. PMID 29254506